CLINICAL TRIAL: NCT02321696
Title: Clinical Comparative Effect of Physiotherapy or Acupuncture Treatment of Lateral Epicondylitis; a Randomized Controlled Pilot Trial
Brief Title: Physiotherapy or Acupuncture for Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Kjersti Storheim, Head of FORMI, Oslo University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1520
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Lateral Epicondylitis
Keywords: physiotherapy; manual therapy; acupuncture; eccentric exercise
MeSH Terms: conditions — Tennis Elbow | interventions — Acupuncture Therapy; Physical Therapy Modalities; Watchful Waiting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture and eccentric exercise (Experimental): Treatment will be performed according to traditional Chinese methods (STRICTA: Standards for reporting interventions in controlled trials of acupunc-ture). Therapists will select points frequently recommended for the treatment of LE. As local point, LI11 and LI10 over the muscular origin of the lateral extensor group of the forearm will be used, and LU5 in the cubical region. LI4 and TE5 will be regional points for pain therapy in the upper limb, GB34 will be used as a distal point for treatment of tendinosis in general, and ST36 for treatment of pain. Needles will be inserted down to the musculature and obtaining De Qi sensation and will remain in situ for 20 min. All patients will receive four treatment sessions; this may be extended to eight depending on patient's pain report and the therapists' clinical evaluation. Maximum treatment period is 4 weeks. Patients will also be instructed in eccentric strength exercises for daily home training from enrolment and 12 weeks forward.
  Interventions: Device: Acupuncture; Other: eccentric exercise
- Physiotherapy and eccentric exercise (Experimental): Manual techniques as gliding mobilization of elbow, therapists are spezialised in manual therapy. At least four treatment sessions will be performed, but depending on the patient's perceived intensity of pain and the therapists' clinical evaluation, a maximum of eight treatment session can be given. All treatment session will be performed during a period of maximum 4 weeks.
  In addition, patients will be instructed in eccentric strength exercises for daily home training from enrolment and 12 weeks forward.
  Interventions: Other: Physiotherapy and eccentric exercise
- Watchful waiting and eccentric exercise (Active Comparator): Patients will be instructed in eccentric strength exercises for daily home training from enrolment and 12 weeks forward.
  Interventions: Other: Watchful waiting and eccentric exercise

INTERVENTIONS:
Device: Acupuncture
  Arms: Acupuncture and eccentric exercise
Other: Physiotherapy and eccentric exercise
  Arms: Physiotherapy and eccentric exercise
Other: Watchful waiting and eccentric exercise
  Arms: Watchful waiting and eccentric exercise
Other: eccentric exercise
  Arms: Acupuncture and eccentric exercise

SUMMARY:
Work-related upper extremity disorders are common problems in working populations in western countries. Lateral epicondylitis (LE) or tennis elbow is the most frequent type of soft tissue syndrome of the elbow, with an annual incidence of four to seven cases per 1000 patients in general practice, and as high as 15 % of workers in highly repetitive hand task industries.

LE is a painful condition, leading to loss of function of the affected limb. Therefore it can have a major impact on the patient's work and personal life. If untreated, it persists for an average of six to 24 months and associated with significant sickness absence in 5 % of affected working-aged adults. The cost is therefore high, both in terms of loss of productivity and health care utilization.

Many treatments have been advocated in the management of LE, possibly implying that much is unknown about its etiology and how it best should be treated. Systematic reviews have failed to draw any firm conclusions as to what treatment is most effective in managing this condition.

Over the past 10 years acupuncture has gained wider acceptance for treating pain, by both clinicians and consumers of health, and there is some evidence suggesting that acupuncture treatment is effective in of acute symptoms in LE. A recent study supports that also elbow manipulation have a short-term relief of acute symptoms in LE, especially when combined with eccentric exercise. Our study will therefore explore the clinical effectiveness of physiotherapy versus acupuncture treatment of LE, compared with watchful waiting.

DETAILED DESCRIPTION:
The study design is three armed and randomized, single blinded. The study aims, in a pilot stydy, to test if physiotherapy or acupuncture treatment of lateral epicondylitis, compared with watchful waiting, is useful means in pain relief for patients with lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Lateral epicondylitis LE (duration > 2 weeks)
* Unilateral localization
* Individuals with average pain of NRS 4 or higher during the last week prior to screening
* Aged between 18 and 67 years
* Written informed consent

Exclusion Criteria:

* Corticosteroid injections during the last 4 weeks
* Diseases of the central or peripheral nervous system
* Inflammatory rheumatic diseases
* Radio-ulna or radio humeral osteoarthritis
* Unwilling to participate

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Elbow pain on Numeric Rating Scale (0-10) | 12 weeks and 1 year
  present, worst and lesser pain during the last week, an average score will be calculated

SECONDARY OUTCOMES:
The disabilities of the arm shoulder and hand (quick-DASH) | 12 weeks and 1 year
  Functional capacity of elbow and arm
Quality of life by EQ-5D | 12 weeks and 1 year
  Quality of life
Sick listing | 12 weeks and 1 year
  Number of days patients are sich listed during the 12 week study period
Patients satisfaction; global perceived effect and satistfaction with treatment | 12 weeks and 1 year
Use of analgesics | 12 weeks and 1 year
Number of treatment sessions | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Wahl, PhD, Study Director — University of Oslo
Locations (1):
- Norsk Idrettsmedisinsk Institutt Ullevål, Oslo, Norway

REFERENCES:
- [Derived] Bostrom K, Maehlum S, Cvancarova Smastuen M, Storheim K. Clinical comparative effectiveness of acupuncture versus manual therapy treatment of lateral epicondylitis: feasibility randomized clinical trial. Pilot Feasibility Stud. 2019 Sep 7;5:110. doi: 10.1186/s40814-019-0490-x. eCollection 2019. PMID 31516727